CLINICAL TRIAL: NCT02892383
Title: Quality of Life in Danish Multiple Myeloma Patients
Brief Title: Quality of Life the Danish Multiple Myeloma Patients
Acronym: QoL-MM
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: Danish Myeloma Study Group (Other)
Responsible Party: Principal Investigator, Lene Kongsgaard Nielsen, Specialist in Haematology, Odense University Hospital
Other Study IDs: QoL-MM_OUH
Record Dates: First submitted 2016-06-14; First posted 2016-09-08 (Estimated); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Quality of Life; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the project is to improve quality of life for multiple myeloma patients in the future.

DETAILED DESCRIPTION:
Multiple myeloma is an incurable malignancy of the bone marrow and the second most common type of haematological cancer. In Denmark, about 320 patients are diagnosed annually with multiple myeloma, and the cancer often affects older people, but 30 % of the patients living with MM are of working age. The prognosis has improved markedly over the last two decades and is expected to improve further.

Systematic monitoring of symptoms, side effects and complications over time outside clinical trials has not been performed yet. Knowledge of the elderly and frail patients´ perspective on the multiple myeloma disease is lacking, and the time after anti-myeloma treatment is left unstudied. A common side effect (up to 55 %) to specific types of anti-myeloma drugs is peripheral neuropathy (nerve injury), which can be temporary or permanent in the form of long-term sequelae of pain and numbness. Information on this side effect from the patients´ perspective is missing.

The design of the project is a prospective, population-based, national, longitudinal survey with retrospective data collection from more Danish registers. We will include 800 previously untreated and relapsed multiple myeloma patients at treatment-demanding disease recruited from all Danish haematological departments. At inclusion, demographic data and patient-related prognostic markers will be obtained. The patients will complete four validated QoL instruments (EORTC QLQ-C30, MY20, CIPN20 and SF12v2) at 13 measuring points over a period of 24 months. The questions are concerning cancer and MM symptoms, peripheral neuropathy, other side effects, quality of life and functional capacity of a social, emotional and physical character.

This project will provide real-time data collection of the symptoms, side effects, complications and quality of life from the general multiple myeloma patients´ perspective during and after anti-myeloma treatment. It will illuminate the reason for the patients´ high loss of working ability. The findings will be integrated in the future Danish National treatment guidelines, and recommendation for rehabilitation in aspects of shared decision making.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated or relapsed multiple myeloma patients AND
* Treatment demanding multiple myeloma disease

Exclusion Criteria:

* Inability to understand the Danish language or
* Psychic or mental illness that prevents the patient from answering the questions in the questionnaires.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Danish multiple myeloma patients
Sampling Method: Non-Probability Sample
Enrollment: 681 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
A longitudinal description of quality of life (QoL) using patient-reported outcomes measurement (PROM) for the general population of multiple myeloma patients. | 24 months
  a. Description of changes in QoL over time

SECONDARY OUTCOMES:
Description of changes in QoL over time, based on PROM for the general population of multiple myeloma patients. | 24 months
  1. To analyse changes in QoL measured by EORTC QLQ-C30 (score 0-100), EORTC QLQ-MY20 (score 0-100) and SF12v2-4-week recall (score 0-100) in relation to disease characteristics:
     * ISS I-III
     * Type/-s of anti-myeloma treatment
     * Side-effects of treatment measured by EORTC QLQ-MY20 (score 0-100) and EORTC QLQ-CIPN20 (score 0-100)
     * Quality of response: IMWG criteria for first and second line treatment
  2. To analyse changes in QoL measured by EORTC QLQ-C30 (score 0-100), EORTC QLQ-MY20 (score 0-100) and SF12v2-4-week-recall (score 0-100) in relation to patient characteristics:
     * Myeloma Frailty score (fit, intermediate-fitness and frail)
     * Karnofsky Performance score scale (0-100%)
     * Charlson comorbidity Index (0-33) and Freiburger comorbidity index (0-3)
Description of the impact of peripheral neuropathy on QoL in the general population of multiple myeloma patients over time, based on PROM. | 24 months
  1. To analyse changes in peripheral neuropathy measured EORTC QLQ-CIPN20 (score 0-100) in relation to
     * Type/-s of anti-myeloma treatment
     * Side effect of treatment measured by EORTC QLQ-MY20 (score 0-100).
     * Quality of response: IMWG criteria for first and second line treatment
  2. To analyse changes in peripheral neuropathy measured by EORTC QLQ-CIPN20 (score 0-100) in relation to - Myeloma frailty score (fitness, intermediate-fitness and frail)
Description of the impact of recalibration response shift for interpretation of data from longitudinal QoL studies using PROM for QoL measurement in the general population of previously untreated multiple myeloma patients. | 9 months
  Recalibration response shift is a change in the patients internal standard of Measurement and will be measured at a then-test interview 9 months after baseline. Then-test is a retrospective pre-test and will capture recalibration response shift and the true change in QoL. For the pre-test, post-test and then-test the EORTC QLQ-C30 (score 0-100), EORTC QLQ-MY20 (score 0-100), EORTC QLQ-CIPN20 (score 0-100) and SF12v2-4-week recall (score 0-100) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Lene Kongsgaard Nielsen, MD, Principal Investigator — Quality of Life Research Centre, Haematological Department, Odense Univsersity Hospital
Locations (10):
- Denmark (10):
  - Sygehus Sønderjylland, Aabenraa
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Sydvestjysk Sygehus, Esbjerg
  - Herlev Hospital, Herlev
  - Hospitalsenheden Vest, Holstebro
  - Odense University Hospital, Odense
  - Sjællands Universitetshospital, Roskilde
  - Vejle Sygehus, Vejle

IPD SHARING:
Plan to Share IPD: Yes
The cohort will be used as historical controls in clinical intervention trials

REFERENCES:
- [Derived] Engelhardt M, Ihorst G, Singh M, Rieth A, Saba G, Pellan M, Lebioda A. Real-World Evaluation of Health-Related Quality of Life in Patients With Multiple Myeloma From Germany. Clin Lymphoma Myeloma Leuk. 2021 Feb;21(2):e160-e175. doi: 10.1016/j.clml.2020.10.002. Epub 2020 Oct 24. PMID 33218965